CLINICAL TRIAL: NCT02243878
Title: StereoTactic Radiotherapy for Wet Age-Related Macular Degeneration (STAR): A Randomised, Double-masked, Sham-controlled, Clinical Trial Comparing Low-voltage X-ray Irradiation With as Needed Ranibizumab, to as Needed Ranibizumab Monotherapy.
Brief Title: Stereotactic Radiotherapy for Wet AMD (STAR)
Acronym: STAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UKCRN ID 18040; ISRCTN12884465 (Registry Identifier: International Standard Randomised Controlled Trial Number(ISRCTN)); EME-Project:12/66/22 (Other Grant/Funding Number: National Institute for Health Research)
Record Dates: First submitted 2014-09-08; First posted 2014-09-18 (Estimated); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Neovascular (Wet) Age-related Macular Degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration | interventions — Radiosurgery; salicylhydroxamic acid; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (treatment) (Experimental): Participants will receive Stereotactic radiotherapy, a 16 Gy dose of radiation, delivered to the macula.
  Participants will receive intravitreal injections of 0.5 mg ranibizumab at baseline, and then administered 'as required' (PRN) up to monthly, if predefined retreatment criteria are met.
  Interventions: Radiation: Stereotactic radiotherapy (16 Gray or Sham); Drug: 0.5 mg ranibizumab
- Arm B (control) (Sham Comparator): Participants will receive a sham treatment.
  Participants will receive intravitreal injections of 0.5 mg ranibizumab at baseline, and then administered 'as required' (PRN) up to monthly, if predefined retreatment criteria are met.
  Interventions: Radiation: Stereotactic radiotherapy (16 Gray or Sham); Drug: 0.5 mg ranibizumab

INTERVENTIONS:
Radiation: Stereotactic radiotherapy (16 Gray or Sham) — Participants will be allocated in a 2:1 ratio to either 16 Gray SRT (IRay, Oraya, Newark,USA) delivered in a single session, or sham SRT.
Drug: 0.5 mg ranibizumab — Both arms will receive intravitreal injections of 0.5 mg ranibizumab at baseline, and then administered 'as required' (PRN) up to monthly, if predefined retreatment criteria are met.
  Other Names: Lucentis®

SUMMARY:
This study investigates the use of radiation to treat wet age-related macular degeneration (AMD). The radiation is delivered using a robotically controlled device that projects overlapping beams of radiation onto the macula, the part of the eye that is affected by wet AMD. Participants will be randomized to receive radiation (stereotactic radiotherapy) or simulated placebo treatment (sham control). They will be followed up regularly for two years, and then again at the end of three and four years for a safety visit. Participants will also receive injections of ranibizumab (Lucentis) into their eye if their wet AMD is active. Ranibizumab is the standard anti-VEGF agent that is used to treat wet AMD. The study aims to determine if stereotactic radiosurgery can maintain vision and reduce the need for such regular anti-VEGF injections.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) leads more people to go blind than all other eye diseases combined. 'Wet' AMD occurs when abnormal new blood vessels grow into the macula. The macula is an area inside the back of the eye, which is tightly packed with the light-sensitive cells that give fine central vision for driving, reading, facial recognition etc. Most patients are treated with repeated injections of ranibizumab (Lucentis), bevacizumab (Avastin) , or aflibercept (Eylea) into the eye (these drugs suppresses the new vessel growth). Unsurprisingly, the need for hospital visits every 1-2 months, and regular injections into the eye, is not favoured by patients.

The proposed study investigates the use of radiation to treat wet AMD. Radiation preferentially damages proliferating cells, such as those forming the abnormal new blood vessels. It has the potential to kill off the abnormal cells, unlike the injections which just suppress the disease.

The radiation is delivered using a robotically controlled device that aims three beams of radiation in through the white of eye, to overlap at the macula. Initial studies of stereotactic radiotherapy (SRT) were promising, and established the best dose of radiation. They showed that radiation has the potential to significantly reduce the need for injections. Each injection costs the National Health Service (NHS) approximately £600, hence the potential cost savings are substantial. For those who respond well, disease activity is reduced, and injections can be eliminated or greatly reduced.

Eye charities have run focus groups of people with wet AMD to help set priorities, and participants identified the burden of treating wet AMD as one of their most pressing concerns, as it greatly restricts their freedom and quality of life. Repeated injections also carry risks of rare but blinding complications, and long term they may possibly lead to other eye diseases such as glaucoma and atrophy of the macula.

The preliminary SRT studies were not designed to determine if the visual outcome was the same, better, or worse than standard injection therapy, and follow up was too short to determine long term risks. A larger study is therefore required to confirm that SRT reduces the number of injections and to determine if the visual outcomes are acceptable. There is also a need for longer term safety monitoring, as radiation damage typically has a delayed onset.

STAR will use ranibizumab as the anti-VEGF agent in both the treatment and control arms. Ranibizumab was chosen over bevacizumab as it is licensed for use in the eye, and at present bevacizumab is used in only a small minority of NHS hospitals, such that the results with bevacizumab may be less generalisable. Bevacizumab may slow recruitment if prospective participants are anxious about swapping to an off label treatment, and preliminary discussions with prospective sites indicated some investigators would prefer to use ranibizumab. Further, ranibizumab was used in the phase II INTREPID study (detailed below), which helps inform the STAR statistical analysis. Aflibercept's mandated dosing in year 1 means it is not possible to determine if radiation reduces the need for anti-VEGF treatment, the primary outcome measure.

Participants will be randomly allocated to dummy SRT (0 Gray dose) or live SRT (16 Gray). Neither the treating doctor nor participant will know if a 0 or 16 Gray dose was given. SRT will be performed in approximately 3 national treatment centres, but 25 NHS recruiting hospitals will refer patients for SRT, and then review them afterwards, treating them with ranibizumab as needed.

Participants will attend for examination monthly for two years. They will then revert to standard NHS care, but with two further study visits - one at the end of year 3 and one at the end of year 4. These two late safety visits are to exclude delayed radiation damage. At the 24 monthly visits participants will have their vision tested on an eye chart, and a laser scan (OCT) of their macula. If the vision drops or the OCT shows disease activity, then they will receive an injection of ranibizumab. Participants will have imaging of the blood vessels in the macula (angiography) at baseline and yearly thereafter for 4 years. The images will be interpreted by an independent, specialist reading centre to quantify the effect of treatment, to study the interaction of radiation and wet AMD, to look for subtle radiation damage, and to subclassify disease to determine who responds best to SRT.

We predict that SRT will produce a similar, or possibly better vision than ranibizumab alone, but with fewer injections. With 411 participants we will have 90% certainty that our results are valid.

Participants will provide feedback using established questionnaires about how acceptable they found SRT, their visual function, and their overall quality of life. Experienced health economists will then look at the cost of treatment in relation to any improvement in quality of life, to see if SRT is cost-effective.

The main outcomes we will monitor are the number of eye injections and visual function on an eye chart, but several other observations will be made. In particular, we will monitor the safety of treatment, any collateral damage caused by radiation, and the interactions between radiation and diseased eye tissue.

If proven to be effective, SRT has the potential to save the NHS money, but more importantly, it may reduce the burden of care faced by more than 250,000 people with wet AMD.

ELIGIBILITY:
Inclusion Criteria

1. Participants must have neovascular AMD in the study eye, for which they have received at least 3 prior intravitreal injections of either bevacizumab (Avastin), aflibercept (Eylea), ranibizumab (Lucentis), or pegaptanib (Macugen).
2. Participants must have received an anti-VEGF injection in the study eye within 3 months prior to enrolment.
3. Participants must require treatment with anti-VEGF therapy at the time of enrolment, due to OCT evidence of subretinal fluid and/or cystoid macular oedema, and have a macular volume that is greater than the 95th percentile of normal for the SD-OCT machines used in the investigational sites.
4. Participants must be at least 50 years of age.

Exclusion Criteria

1. Disciform scarring that involves the fovea, in the study eye.
2. Visual acuity worse than 6/96 (24 ETDRS letters) in the study eye.
3. Lesion size greater than 4 mm in greatest linear dimension, or greater than 2 mm from the centre of the fovea to the furthest point on the lesion perimeter.
4. An axial length of less than 20 mm, or greater than 26 mm, in the study eye.
5. Contraindication or sensitivity to contact lens application, including recurrent corneal erosions, in the study eye.
6. Type 1 or Type 2 diabetes mellitus.
7. Retinopathy in the study eye.
8. Prior or current therapies in the study eye for age-related macular degeneration, other than anti-VEGF agents, including submacular surgery, subfoveal thermal laser photocoagulation, photodynamic therapy (PDT), or transpupillary thermotherapy (TTT).
9. Presence of an intravitreal device in the study eye.
10. Previous radiation therapy to the study eye, head, or neck with the exception of radio-iodine treatment for hyperthyroidism, epimacular brachytherapy to the non-study eye, or Oraya SRT to the non-study eye.
11. Inadequate pupillary dilation or significant media opacities in the study eye, including cataract, which may interfere with visual acuity testing, the clinical evaluation of the posterior segment, or fundus imaging.
12. Study eyes with CNV due to causes other than AMD, including presumed ocular histoplasmosis syndrome (POH), angioid streaks, multifocal choroiditis, choroidal rupture, and pathological myopia (greater than 8 Dioptres spherical equivalent). Participants with retinal angiomatous proliferation (RAP) or idiopathic polypoidal choroidal vasculopathy (IPCV) are not excluded.
13. Known allergy to intravenous fluorescein, ICG or intravitreal ranibizumab.
14. Intraocular surgery or laser-assisted in situ keratomileusis (LASIK) in the study eye within 12 weeks prior to enrolment.
15. Prior pars plana vitrectomy in the study eye.
16. Current participation in another interventional clinical trial, or participation in such a clinical trial within the last six months.
17. Unwilling, unable, or unlikely to return for scheduled follow-up for the duration of the trial.
18. Women who are pregnant at the time of radiotherapy.
19. Participants with an implantable cardioverter defibrillator (ICD) or pacemaker implant (or any implanted device) where the device labelling specifically contraindicates patients undergoing X-ray.
20. Any other condition, which in the judgment of the investigator, would prevent the participant from granting informed consent or completing the study, such as dementia, and mental illness (including generalized anxiety disorder and claustrophobia).

Ages: 50 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Estimated)
Dates: Start 2014-12; Primary Completion 2021-12 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Number of as required (prn) ranibizumab injections during the first 24 months | 24 months
  Monitor the number of eye injections

SECONDARY OUTCOMES:
Mean Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity (VA) at 24 months. | 24 months
  Measure the visual function on an eye chart

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Jackson, PhD FRCOphth, Principal Investigator — King's College Hospital NHS Trust
Locations (30):
- United Kingdom (30):
  - Bristol Eye Hospital, Bristol, Bristol
  - Hinchingbrooke Hospital, Huntingdon, Cambridgeshire
  - The Princess Alexandra Hospital, Harlow, Essex
  - Maidstone Hospital, Maidstone, Kent
  - Ashford William Harvey Hospital, Willesborough, Kent
  - James Paget University Hospital, Great Yarmouth, Norfolk
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - Frimley Park Hospital, Frimley, Surrey
  - Stoke Mandeville Hospital, Aylesbury
  - Heart Of England NHS Foundation Trust, Birmingham
  - Royal Blackburn Hospital, Blackburn
  - Sussex Eye Hospital, Brighton
  - Addenbrooke's Hospital, Cambridge
  - Essex County Hospital, Colchester
  - Leighton Hospital, Crewe
  - Royal Derby Hospital, Derby
  - Dorset County Hospital, Dorchester
  - Calderdale Royal Hospital, Halifax
  - Whipps Cross Hospital, Leytonstone
  - Lincoln Country Hospital, Lincoln
  - Central Middlesex Hospital, London
  - King's College Hospital NHS Foundation Trust, London
  - Epsom and St. Helier Hospital, London
  - Manchester Royal Eye Hospital, Manchester
  - Norfolk & Norwich University Hospital, Norwich
  - Queen's Hospital, Romford
  - Salisbury District Hospital, Salisbury
  - Hillingdon Hospital, Uxbridge
  - New Cross Hospital, Wolverhampton
  - Yeovil District Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jackson TL, Desai R, Wafa HA, Wang Y, Peacock J, Peto T, Chakravarthy U, Dakin H, Wordsworth S, Lewis C, Clinch P, Ramazzotto L, Neffendorf JE, Lee CN, O'Sullivan JM, Reeves BC; STAR study group. Stereotactic radiotherapy for neovascular age-related macular degeneration (STAR): a pivotal, randomised, double-masked, sham-controlled device trial. Lancet. 2024 Jul 6;404(10447):44-54. doi: 10.1016/S0140-6736(24)00687-1. Epub 2024 Jun 11. PMID 38876132
- [Derived] Neffendorf JE, Desai R, Wang Y, Kelly J, Murphy C, Reeves BC, Chakravarthy U, Wordsworth S, Lewis C, Peacock J, Uddin S, O'Sullivan JM, Jackson TL. StereoTactic radiotherapy for wet Age-Related macular degeneration (STAR): study protocol for a randomised controlled clinical trial. Trials. 2016 Nov 24;17(1):560. doi: 10.1186/s13063-016-1676-7. PMID 27881184